CLINICAL TRIAL: NCT01293799
Title: Prevention of Peritonitis in Patients With Peritoneal Dialysis - Effects of Regular Follow-up of Patients´ Theoretical Knowledge and Practical Skills With Focus on Infection Prophylaxis
Brief Title: Prevention of Peritonitis in Peritoneal Dialysis
Acronym: PEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Sykehuset Innlandet HF (Other); Tampere University Hospital (Other); Pauls Stradins Clinical University Hospital (Other); Tartu University Hospital (Other); Karolinska Institutet (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Susanne Ljungman, professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 590-09
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Kidney Failure, Chronic; Peritoneal Dialysis-associated Peritonitis; Dialysis Capd Infection
Keywords: Randomized; Peritoneal dialysis; Peritonitis; Primary prevention; Quality control; Self care; Kidney failure, chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis

STUDY DESIGN:
Intervention Model Description: A non-commercial, physician-initiated, randomized, controlled, open-label, parallel-group, multicenter clinical trial. The participants were randomly assigned to either retraining with testing of their peritoneal dialysis knowledge (the retraining group) or to usual care (the control group).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The retraining group (Experimental): The intervention in the retraining group consists of regular tests of the patients´ theoretical and practical skills regarding peritoneal dialysis. The test goals should be passed. If not, retraining will be given if needed til the goals are reached. The peritonitis rate in this group will be compared with that of the control group.
  Interventions: Behavioral: Retraining
- Control group (No Intervention): Patients randomised to the control group will be treated according to the routines of the clinic.

INTERVENTIONS:
Behavioral: Retraining — Testing of the patients´ knowledge and retraining will be given if needed
  Arms: The retraining group

SUMMARY:
BACKGROUND: Peritonitis remains a significant problem in peritoneal dialysis (PD). It is the leading cause of technique failure, and contributes to mortality. The incidence is highest during the first year of treatment. Non-compliance with the PD protocol is shown to be an important risk factor for peritonitis. Reinforcement of knowledge and ability to perform PD therefore appears to be a possible way to reduce the incidence of peritonitis. This will be studied in The PEritonitis Prevention Study (PEPS).

METHODS: The objective of this randomized, multi-centre investigation, which will include 750 new PD patients who can perform (PD) without assistance, is to evaluate if regular retraining can reduce the incidence of peritonitis, the technique-failure rate, and the hospitalisation days due to peritonitis compared with regular follow-up regimen. Patients in the intervention group will be tested by a PD-technique test and a questionnaire at regular intervals after PD-start and after every peritonitis episode with focus on infection prophylaxis. If needed, they will be retrained. The control group will be treated according to the routine of the center.

The study is ongoing in Denmark, Norway, Sweden, Finland, Estonia, Latvia, the Netherlands, and the United Kingdom (UK). The study will go on for 6 years.

DETAILED DESCRIPTION:
BACKGROUND See above.

AIMS The primary aim of this trial is to study if regular follow-up of PD patients with testing of their theoretical and practical knowledge (hereafter called "new type of follow-up") can reduce the time to first peritonitis episode. Secondary aims were to study if the new type of follow-up could reduce the incidence of peritonitis, the technique failure rate related to peritonitis, and the time of hospitalization related to peritonitis compared to a routine regimen. For specific aims, see "Outcome measures" below. A further aim was to study risk factors for peritonitis.

PATIENTS AND METHODS The study is a randomized, multi-centre investigation intending to enclose 750 new PD patients in Sweden, Denmark, Norway, Finland, Estonia, Latvia, the Netherlands, and the United Kingdom. Inclusion was finished on December 31, 2014. The study will go on until the last included patient has taken part of the study for one year. The study will thus be terminated on December 31, 2015.

The study includes a retraining group and a control group. The intervention in the retraining group consists of regular testing of theoretical and practical knowledge regarding PD with focus on infection prophylaxis including retraining if needed until the test goals are reached. The control group will be treated according to the routines of the center. Peritonitis is defined according to International Society for Peritoneal Dialysis (SPD) guidelines (Peritoneal Dialysis International 2005;25:107-131)

The baseline PD training will be the same at all participating centres and follow international recommendations. In addition, fluorescent alcohol and a UV lamp will be used to control the result of hand disinfection in all patients once during the initial PD training. Thereafter this method will only be used in the retraining group..

In the retraining group, the knowledge from the basal training will be tested at 1, 3, 6, and 12 months after PD start, every sixth month thereafter, and after every episode of peritonitis. Such testing will also be performed at restart of PD and includes two types of tests:

1. The patient will fill in a questionnaire with theoretical and practical questions with focus on infection and infection prophylaxis during PD treatment. Goal: At least 80% of the questions should be correct. If the goal is not reached, further training will be given until the goal is reached.
2. The patient will perform a practical test including hand disinfection, PD exchange technique, and exit-site care. Hand disinfection skills will be controlled with the help of fluorescent alcohol and a UV lamp. Goal: All steps of the practical test should be correctly performed. If not, further training will be given until the goal is reached.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to perform PD without assistance
* Age 18 years old or more

Exclusion Criteria:

* Previous PD-treatment less than 2 years ago
* Peritonitis before inclusion
* Active malignancy
* Participation in other studies during the study period which may affect outcome of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Ljungman, Prof. emer., Study Director — Department of Nephrology, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Department of Nephrology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on January 18th, 2010 and ended on December 31st, 2014. The recruitment time was prolonged from planned two years to five years. Of the 713 initially included subjects, only 671 met the inclusion criteria. Of the 671 randomized subjects, 331 were assigned to the Control group and 340 to the Follow-up group.
Groups:
- The Retraining Group: 340 patients were allocated to the retraining group.
- Control Group: 331 subjects were allocated to the Control group.
Period: Overall Study
Arm/Group | The Retraining Group | Control Group
Started | 340 | 331
First Peritonitis Episode | 102 (102 of the participants in this group suffered at least one peritonitis episode) | 121 (121 of the participants suffered in this group at least one peritonitis episode.)
Completed | 67 | 86
Not Completed | 273 | 245
Not completed — Kidney transplantation | 109 | 96
Not completed — Transfer to hemodialysis | 70 | 90
Not completed — Death | 27 | 29
Not completed — Transfer to assisted PD | 24 | 18
Not completed — Withdrawal by Subject | 26 | 0
Not completed — Investigator decision | 5 | 2
Not completed — Kidney function improved | 6 | 7
Not completed — Other causes | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- The Retraining Group: The intervention in the retraining group consisted of tests at the study visits of the patients´ theoretical and practical skills regarding peritoneal dialysis If the test goals were not passed, retraining was given until the goals were reached. The peritonitis rate in this group will be compared with that of the control group.
- Control Group: Patients randomised to the control group were treated according to the routines of the clinic.
- Total: Total of all reporting groups
Arm/Group | The Retraining Group | Control Group | Total
Number analyzed (Participants) | 340 | 331 | 671
Age, Continuous [Median (Full Range); unit: Years] | 64 [19 to 87] | 62 [19 to 88] | 62 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 114 | 225
  Male | 229 | 217 | 446
Region of Enrollment [Number; unit: participants]
  Sweden | 191 | 192 | 383
  Latvia | 25 | 25 | 50
  Netherlands | 25 | 26 | 51
  Denmark | 32 | 27 | 59
  Estonia | 11 | 9 | 20
  Norway | 30 | 26 | 56
  Finland | 22 | 22 | 44
  United Kingdom | 4 | 4 | 8
Age 65 years or more [Count of Participants; unit: Participants] | 164 | 144 | 308
Body weight [Mean (Standard Deviation); unit: Kg] | 77 (15) | 79 (16) | 78 (15)
Body mass index [Mean (Standard Deviation); unit: Kg/m2] | 26 (4) | 26 (4) | 26 (4)
Primary cause of end-stage kidney disease [Count of Participants; unit: Participants]
  Diabetic nephropathy | 63 | 87 | 150
  Glomerulonephritis | 87 | 87 | 174
  Tubulointerstitial nephritis | 17 | 17 | 34
  Polycystic kidney disease | 40 | 29 | 69
  Ischemic kidney kisease | 1 | 1 | 2
  Nephrosclerosis/Hypertension | 78 | 66 | 144
  Other diagnosis | 38 | 26 | 64
  Unknown cause | 16 | 18 | 34
Comorbidity [Number; unit: participants]
  Ischemic heart disease | 60 | 62 | 122
  Peripheral vascular disease and stroke | 39 | 27 | 66
  Left ventricular dysfunction | 37 | 34 | 71
  Diabetes (comorbidity or main cause of kidney failure) | 88 | 111 | 199
  Collagen vascular disease | 20 | 10 | 30
  Other significant pathology | 42 | 30 | 72
Karnofsky performance scale for measurement of functional status [Median (Full Range); unit: Score] — Scores:
  100 Normal no complaints; no evidence of disease.
  90 Able to carry on normal activity; minor signs or symptoms of disease
  80 Normal activity with effort; some signs or symptoms of disease.
  70 Cares for self; unable to carry on normal activity or to do active work.
  60 Requires occasional assistance; but able to care for most of his/her personal needs.
  50 Requires considerable assistance and frequent medical care.
  40 Disabled; requires special care and assistance.
  30 Severely disabled; hospital admission indicated although death not imminent.
  Score | 90 [80 to 95] | 90 [80 to 90] | 90 [80 to 90]
Social factors [Count of Participants; unit: Participants]
  Visual impairment with reading problems | 17 | 28 | 45
  Impaired hand function | 23 | 21 | 44
  Working full or part time | 103 | 102 | 205
  Retired | 184 | 169 | 353
  Living alone | 91 | 77 | 168
  Need for translation/interpreter | 9 | 13 | 22
  Current smoking | 34 | 39 | 73
Serum creatinine (at PD start) [Mean (Standard Deviation); unit: Micromol/L] — Baseline laboratory tests were performed just before the start of peritoneal dialysis
  Micromol/L | 640 (234) | 650 (208) | 645 (222)
Serum urea (at PD start) [Mean (Standard Deviation); unit: mmol/L] | 28 (9) | 28 (9) | 28 (9)
Serum albumin (at PD start) [Mean (Standard Deviation); unit: g/L] — Population: Data was missing for one subject in the Retraining group and 3 subjects in the Control group.
  g/L
    number analyzed (Participants) | 339 | 328 | 667
    (all) | 34 (6) | 34 (6) | 34 (6)
Serum albumin < 35 g/L (at PD start) [Count of Participants; unit: Participants] — Population: Data was missing for one individual in the Retraining group and 3 individuals in the Control group.
  Participants
    number analyzed (Participants) | 339 | 328 | 667
    (all) | 169 | 169 | 338
Hemoglobin (at PD start) [Mean (Standard Deviation); unit: mmol/L] — Population: Data was missing for one subject in the Retraining group.
  mmol/L
    number analyzed (Participants) | 339 | 331 | 670
    (all) | 110 (14) | 111 (12) | 111 (13)
C-reactive protein [Median (Inter-Quartile Range); unit: g/L] — C-reactive protein analyzed is normally < 3 g/L Population: Data was missing for 2 subjects in the Retraining group and 6 subjects in the Control group.
  g/L
    number analyzed (Participants) | 338 | 325 | 663
    (all) | 3.0 [1.5 to 8.0] | 3.0 [2.0 to 9.0] | 3.0 [2.0 to 9.0]
Medication [Count of Participants; unit: Participants]
  Corticosteroid drug | 44 | 43 | 87
  Other cytotoxic drug | 27 | 25 | 52
  No steroid or other cytotoxic drug medication | 269 | 263 | 532
Participants from centers treating nasal carriers of S. aureus with nasal antibiotics [Count of Participants; unit: Participants] | 73 | 68 | 141
Participants from centers routinely using topical antibiotic cream on catheter exit site [Count of Participants; unit: Participants] | 38 | 34 | 72
Antibiotic prophylaxis before PD catheter insertion [Count of Participants; unit: Participants] | 305 | 305 | 610
Type of PD start [Count of Participants; unit: Participants]
  Planned | 300 | 278 | 578
  Acute | 40 | 53 | 93
PD catheter characteristics [Count of Participants; unit: Participants]
  Straight | 78 | 76 | 154
  Coiled | 262 | 255 | 517
PD modality at PD start [Count of Participants; unit: Participants] — CAPD = Continuous ambulatory peritoneal dialysis APD = Automated peritoneal dialysis
  Participants
    CAPD | 278 | 262 | 540
    APD | 62 | 69 | 131
Help needed with exit-site care [Count of Participants; unit: Participants] — Exit-site = The place where the peritoneal dialysis catheter comes out of the abdominal skin.
  Participants | 79 | 84 | 163

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Dialysis-associated Peritonitis Episode in the Retraining Group and the Control Group
Description: Time (days) after the date of randomization to the date of the first peritonitis episode was calculated for each participant. The cumulative time without peritonitis using the Cox regression model from which unadjusted hazard ratios were calculated. Actuarial survival curves showing proportions of peritonitis-free participants over time in the two groups were estimated by means of the Kaplan-Meier method. Log rank follow-up was used to compare the survival curves. Patients who stopped PD treatment due to causes other than peritonitis were managed according to the intention-to-treat principle.
Time Frame: Participants were followed from 1 month after PD start (time of randomization) up to a maximum of 36 months after start of peritoneal dialysis, i.e. to maximally 35 months after randomization. Time to first peritonitis was calculated for each participant.
Population: A number of 671 new patients with peritoneal dialysis (PD), peritonitis-free, aged 18 years or more, and able to perform PD without assistance were randomized to a control group and a retraining group. Participant who stopped PD treatment due to causes other than peritonitis were managed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: Days to first peritonitis episode
Groups:
- The Retraining Group: The intervention in the retraining group consists of regular tests of the patients´ theoretical and practical skills regarding peritoneal dialysis. The test goals should be passed. If not, retraining will be given if needed til the goals are reached. The peritonitis rate in this group will be compared with that of the control group.
  Follow-up of PD patients´ theoretical and practical skills: Testing of patients knowledge and retraining if needed
Arm/Group | The Retraining Group | Control Group
Number analyzed (Participants) | 340 | 331
Days to first peritonitis episode | 381 [154 to 555] | 368 [161 to 617]
Statistical Analysis 1: Comparison: The Retraining Group vs Control Group; Time to the first peritonitis episode was analyzed as the cumulative time without peritonitis (peritonitis-free survival) using the Cox proportional hazards regression model from which unadjusted hazard ratios (HRs) were calculated. Actuarial survival curves showing proportions of of peritonitis-free participants over time in the two groups were estimated by means of the Kaplan-Meier method. Log-rank follow-up was used to compare the two peritonitis-free survival curves; Test type: Superiority — Patients who stopped PD treatment due to causes other than peritonitis were managed according to the intention-to-treat principle. Patients were censored when the PD treatment was stopped; p = 0.51, Log Rank — The threshold for statistical significance was P = 0.05; Log-rank follow-up was used to compare the peritonitis-free survival curves in the two arms; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.71 to 1.19] — Hazard ratio was the ratio between the hazard rate of the retraining group (nominator) and the hazard rate of the control group (denominator)

2. Secondary Outcome: Incidence of a First Dialysis-associated Peritonitis Episode in the Control and the Retraining Group
Description: The incidence of a first peritonitis episode is expressed as the mean rate of a first peritonitis per patient year (event rate) with 95% confidence interval.
Time Frame: The participants were followed from 1 month after PD start (time of randomization) up to a maximum of 36 months after start of peritoneal dialysis, i.e. to maximally 35 months after randomization. The time in study was calculated for each participant
Population: 671 new patients with peritoneal dialysis, peritonitis-free, aged 18 year or more, and able to perform peritoneal dialysis without assistance were randomized to a control group or a follow-up group and followed up to 36 months after start of peritoneal dialysis. The time (patient-years) in the study to the first peritonitis episode was calculated for for each participant.
Measure: Mean (95% Confidence Interval); unit: Peritonitis events per patient-year
Groups:
- The Retraining Group: Number of individuals allocated to the Retraining group
- Control Group: Number of individuals allocated to the Control group
Arm/Group | The Retraining Group | Control Group
Number analyzed (Participants) | 340 | 331
Peritonitis events per patient-year | 0.29 [0.23 to 0.35] | 0.31 [0.26 to 0.37]
Statistical Analysis 1: Comparison: The Retraining Group vs Control Group; Test type: Other — The number of peritonitis events between the two groups was tested by assuming a Poisson distribution of the number of events per follow-up time, log (follow-up time) as offset time, by using generalized linear models; p = 0.51, Generalized linear methods — P-value <0.05 is regarded as significant; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.70 to 1.19] — In calculation of the Risk Ratio, data for the Retraining group represents the nominator and data for the Control group represents the denominator

3. Secondary Outcome: Incidence of All Peritonitis Episodes in the Control Group and the Retraining Group
Description: The incidence of peritonitis episodes is expressed as the mean rate of peritonitis per patient year (event rate) with 95% confidence interval.
Time Frame: The participants were followed from 1 month after PD start (time of randomization) up to 36 months after start of peritoneal dialysis, The time (days) of participation in the study was calculated for each participant.
Population: 671 new patients with peritoneal dialysis, peritonitis-free, aged 18 year or more, and able to perform peritoneal dialysis without assistance were randomized to a control group or a follow-up group and followed up to 36 months after start of peritoneal dialysis.
Measure: Mean (95% Confidence Interval); unit: Peritonitis event rate per patient year
Arm/Group | Control Group | The Retraining Group
Number analyzed (Participants) | 331 | 340
Peritonitis event rate per patient year | 0.36 [0.31 to 0.41] | 0.33 [0.28 to 0.39]
Statistical Analysis 1: Comparison: Control Group vs The Retraining Group; Test type: Other — The number of recurrent peritonitis events between the two groups was tested by assuming a Poisson distribution of the number of events per follow-up time, log (follow-up time) as offset time, by using generalized linear models; p = 0.54, Generalized linear methods — P-value <0.05 was significant; The analysis includes all peritonitis events in the study; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.75 to 1.16] — In the calculation of the relative risk, data for the retraining group represents the nominator and data for the control group represents the denominator

4. Other Pre Specified Outcome: Analysis of Age in Association With Time to First Peritonitis Episode in the Whole Study Group
Description: The association of baseline variables (at PD start) was studied in the whole study group. Age was recorded at baseline. Data were collected at baseline except for medication, PD modality (CAPD/APD, continuous ambulatory PD/automatic PD), number of PD bags and volume of dialysis fluid used per day, and if help with exit-site care was needed. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: Participants were followed from 1 month after PD start (time of randomization) up to a maximum of 36 months after start of peritoneal dialysis. The time (days) to the first peritonitis episode was calculated for each participant.
Population: 671 new patients with peritoneal dialysis (PD), peritonitis-free, aged 18 years or more, and able to perform PD without assistance were randomized to a control group and a retraining group. We decided to perform the analysis of factors associated with time to first peritonitis in the two groups together, since the possibility to find such associations is likely to be greater in a larger than in a smaller group.
Measure: Median (Full Range); unit: Age, years (See statistical analysis 1)
Groups:
- The Control Group: Patients randomised to the control group will be treated according to the routines of the clinic.
- The Whole Study Group: The Retraining Group and The Control Group together.
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Age, years (See statistical analysis 1) | 64 [19 to 87] | 62 [19 to 88] | 62 [19 to 88]
Statistical Analysis 1: Comparison: The Whole Study Group; The association of age and time to first peritonitis episode is analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other — The association of factors associated with time to first peritonitis was analysed using the Cox proportional hazard regression model. Subjects were censored for various reasons to leave the study. Univariable Cox regression was used to identify factors associated with with time to first peritonitis episode. Multivariable Cox regression was performed using the backward elimination procedure, stopping when all remaining factors were significant at p < 0.05; p = 0.0052, Regression, Cox — Unit of measure: Age (hazard ratio per 10 years). The threshold for statistical significance was P = 0.05; The association of a age (HR per 10 years) and time to first peritonitis episode by univariable Cox regression; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.04 to 1.27]
Statistical Analysis 2: Comparison: The Whole Study Group; Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode (see statistical analysis 1). Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.0041, Regression, Cox — Unit of measure: Age (hazard ratio per 10 years) and time to first peritonitis episode by multivariable Cox regression. The threshold for statistical significance was P = 005; Multivariable Cox regression; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [1.05 to 1.29]

5. Other Pre Specified Outcome: Analysis of "Gender" in Association With Time to First Peritonitis Episode in the Whole Study Group
Description: Outcome data for the baseline variable "Gender" is presented. The association of baseline variables (at PD start) or time-updated variables with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  Male participants | 229 | 217 | 446
  Female participants | 111 | 114 | 225
Statistical Analysis 1: Comparison: The Whole Study Group; The association of gender (male vs. female) and time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.13, Regression, Cox — Unit of measure: Gender (male vs. female). P <0.05 is regarded as statistically significant; Univariable Cox regression was used; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.93 to 1.66]

6. Other Pre Specified Outcome: Analysis of "Body Weight" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for body weight at PD start is presented. The association of baseline variables (at PD start) or time-updated variables with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Kg | 77 (15) | 79 (16) | 78 (15)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of body weight (HR per 10 kg) with time to first peritonitis episode was analysed by univariable Cox regression (Statistical analysis 1) and multivariable Cox regression (Statistical analysis 2); Test type: Other — The association of factors associated with time to first peritonitis was analysed using the Cox proportional hazard regression model. Subjects were censored for various reasons to leave the study. Univariable Cox regression was used to identify factors associated with with time to first peritonitis episode; p = 0.0068, Regression, Cox — Unit of measure: Body weight (hazard ratio per 10 kg). The threshold for statistical significance was P = 0.05; Univariable Cox regression was used; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [1.03 to 1.21]
Statistical Analysis 2: Comparison: The Whole Study Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.03, Regression, Cox — Unit of measure: Body weight (hazard ratio per 10 kg). P < 0.05 is considered significant; Multivariable Cox regression; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [1.01 to 1.19]

7. Other Pre Specified Outcome: Analysis of "Body Mass Index" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for body mass index at PD start is presented. The association of baseline variables (at PD start) or time-updated variables with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: 671 new patients with peritoneal dialysis (PD), peritonitis-free, aged 18 years or more, and able to perform PD without assistance were randomized to a control group and a retraining group. We decided to perform the analysis of factors associated with time to first peritonitis episode in the two groups together, since the possibility to find such associations is likely to be greater in a larger than in a smaller group.
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Kg/m2 | 26 (4) | 26 (4) | 26 (4)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Diabetic nephropathy" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.012, Regression, Cox — Unit of measure: Body mass index (hazard ratio per 5 kg/m2). P < 0,05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [1.04 to 1.38]

8. Other Pre Specified Outcome: Analysis of "Diabetic Nephropathy" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Diabetic nephropathy" as primary cause of kidney failure are presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 63 | 87 | 150
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Diabetic nephropathy" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.56, Regression, Cox — Unit of measure: Diabetic nephropathy as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.66 to 1.25]

9. Other Pre Specified Outcome: Analysis of "Glomerulonephritis" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Glomerulonephritis" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 87 | 87 | 174
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Glomerulonephritis" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.74, Regression, Cox — Unit of measure: Glomerulonephritis as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.78 to 1.42]

10. Other Pre Specified Outcome: Analysis of "Tubulointerstitial Nephritis" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Tubulointerstitial nephritis" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 17 | 17 | 34
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Tubulointerstitial Nephritis" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.42, Regression, Cox — Unit of measure: Tubulointerstitial nephritis as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.73 to 2.15]

11. Other Pre Specified Outcome: Analysis of "Polycystic Kidney Disease" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Polycystic kidney disease" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 40 | 29 | 69
Statistical Analysis 1: Comparison: The Whole Study Group; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.038, Regression, Cox — Unit of measure: Polycystic kidney disease as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Cox regression; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.33 to 0.97]

12. Other Pre Specified Outcome: Analysis of "Ischemic Kidney Disease" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Ischemic kidney disease" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 1 | 1 | 2
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Ischemic kidney disease" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.52, Regression, Cox — Unit of measure: Ischemic kidney disease as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.92, 95% CI 2-sided [0.27 to 13.68]

13. Other Pre Specified Outcome: Analysis of "Nephrosclerosis/Hypertension" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Nephrosclerosis/hypertension" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 78 | 66 | 144
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Nephrosclerosis/Hypertension" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.13, Regression, Cox — Unit of measure: Nephrosclerosis/Hypertension as primary cause of kidney failure vs. all other causes. P < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.93 to 1.71]

14. Other Pre Specified Outcome: Analysis of "Other Diagnosis" as Primary Cause of Kidney Failure in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Other diagnosis" as primary cause of kidney failure is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 38 | 26 | 64
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Other Diagnosis" as primary cause of kidney failure (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.71, Regression, Cox — Unit of measure: "Other Diagnosis as primary cause of kidney failure" vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.58 to 1.45]

15. Other Pre Specified Outcome: Analysis of "Unknown Primary Cause of Kidney Failure" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Outcome data for the baseline variable "Unknown primary cause of kidney failure" as primary cause of kidney failure are presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 16 | 18 | 34
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Unknown Primary Cause of Kidney Failure" as primary cause of kidney failure with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.89, Regression, Cox — Unit of measure: Unknown cause as primary cause of kidney failure vs. all other causes. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.57 to 1.91]

16. Other Pre Specified Outcome: Analysis of "Comorbidity" (According to Stoke Comorbidity Score) in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Comorbidity" in association with time to first peritonitis episode is presented. The Stoke grading system of cardiovascular comorbidity was used to reflect the comorbid burden. Comorbidity was graded "0" when absent, "1" when 1 or 2, and "2" when 3 or more conditions were present.
  The association of baseline variables (at PD start) or time-updated variables with time to first was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  Stoke score 0 (No comorbidity) | 193 | 202 | 395
  Stoke score 1-2 (1-2 comorbidities) | 128 | 117 | 245
  Stoke Score > 2 (More than 2 comorbidities) | 19 | 12 | 31
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Comorbidity" according to Stoke comorbidity score with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.28, Regression, Cox — Unit of measure: Comorbidity at PD start according to Stoke comorbidity score (1-2 vs. 0) i.e. 1-2 comorbidities vs. no comorbidity. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.88 to 1.53]
Statistical Analysis 2: Comparison: The Whole Study Group; [analysis description as in outcome 16, analysis 1]; Test type: Other; p = 0.44, Regression, Cox — Unit of measure: Comorbidity at PD start according to Stoke comorbidity score (>2 vs. 0) i.e. more than 2 comorbidities vs. no comorbidity. P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.68 to 2.45]

17. Other Pre Specified Outcome: Analysis of "Ischemic Heart Disease" as Comorbidity in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Ischemic heart disease" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 60 | 62 | 122
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Ischemic Heart Disease" as Comorbidity with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.07, Regression, Cox — Unit of measure: Ischemic heart disease as comorbidity at baseline (yes vs. no). P < 0.5 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.97 to 1.87]

18. Other Pre Specified Outcome: Analysis of "Peripheral Vascular Disease or Stroke" as Comorbidity in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Peripheral vascular disease or stroke" (yes vs. no) in association with time to first peritonitis episode is presented. Peripheral vascular disease or stroke"" includes distal aortic, renovascular, and cerebrovascular disease as well as symptomatic disease in these vascular territories e.g. cerebrovascular accident, claudication, amputation or significant stenosis >50% on vascular imaging or Doppler ultrasound. The association of baseline variables with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 39 | 27 | 66
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Peripheral Vascular Disease or Stroke" as Comorbidity with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.80, Regression, Cox — Unit of measure: "Peripheral vascular disease or stroke" as comorbidity at PD start (yes vs. no). P-value <0.05 regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.69 to 1.63]

19. Other Pre Specified Outcome: Analysis of "Left Ventricular Dysfunction" as Comorbidity in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Left ventricular dysfunction" (yes vs. no) in association with time to first peritonitis episode is presented. Left ventricular dysfunction includes clinical evidence of pulmonary oedema not attributable to errors in fluid balance or moderate to severe left ventricular dysfunction on echocardiography, or clinical signs of symptomatic moderate to severe heart failure. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 37 | 34 | 71
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Left ventricular dysfunction as comorbidity" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.53, Regression, Cox — Unit of measure: "Left ventricular dysfunction as comorbidity" (yes vs. no). P-value <0.05 is significant; Univariable Cox regression; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.75 to 1.77]

20. Other Pre Specified Outcome: Analysis of "Diabetes Mellitus as Comorbidity" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Diabetes mellitus as comorbidity" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 25 | 24 | 49
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Diabetes Mellitus as Comorbidity" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.099, Regression, Cox — Unit of measure: "Diabetes Mellitus as Comorbidity" (yes vs. no). P-value < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.93 to 2.22]

21. Other Pre Specified Outcome: Analysis of "System Collagen Vascular Disease" as Comorbidity in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "System collagen vascular disease" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 20 | 10 | 30
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "System Collagen Vascular Disease" as Comorbidity" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.22, Regression, Cox — Unit of measure: "System Collagen Vascular Disease" as Comorbidity" (yes vs. no). P-value <0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.29 to 1.32]

22. Other Pre Specified Outcome: Analysis of "Other Significant Pathology" as Comorbidity in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Other significant pathology" (yes vs. no) in association with time to first peritonitis episode is presented. Other significant pathology includes diseases like severe chronic obstructive airway disease, liver cirrhosis, psychotic illness, and severe osteoarthritis. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 42 | 30 | 72
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Other Significant Pathology as Comorbidity" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.79, Regression, Cox — Unit of measure: "Other Significant Pathology" as Comorbidity (yes vs. no). P < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.61 to 1.46]

23. Other Pre Specified Outcome: Analysis of "Diabetes Mellitus as Comorbidity or Main Cause of Kidney Failure" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Diabetes mellitus as comorbidity or main cause of kidney failure" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 88 | 111 | 199
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Diabetes Mellitus as Comorbidity or Main Cause of Kidney Failure" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.69, Regression, Cox — Unit of measure: "Diabetes Mellitus as Comorbidity or Main Cause of Kidney Failure" (yes vs. no". P-value < 0.05 is regarded as significantly significant; Univariable Cox regression; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.80 to 1.40]

24. Other Pre Specified Outcome: Analysis of "Previous Kidney Replacement Therapy" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Previous kidney replacement therapy" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 68 | 61 | 129
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Previous Kidney Replacement Therapy" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.86, Regression, Cox — Unit of measure: "Previous Kidney Replacement Therapy" (yes vs. no). P-value < 0.05 is regarded as significant; Univariable Cox regression; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.74 to 1.42]

25. Other Pre Specified Outcome: Analysis of "Functional Status (Karnofsky Score)" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Functional status (Karnofsky score)" in association with time to first peritonitis episode in the whole study group is presented. Functional status was estimated using the Karnofsky Performance Scale with scores from 100 (Normal, no complains, no evidence of disease) to 0 (dead). 90 = Able to carry on normal activity, minor signs or symptoms of disease. 80 = Normal activity with effort, some signs or symptoms of disease. 70 = Cares for self, unable to carry on normal activity or do active work. 60 = Requires occasional assistance, but able to to care for most of her/his needs. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Karnofsky score numbers
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Karnofsky score numbers | 90 [80 to 95] | 90 [80 to 90] | 90 [80 to 90]
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Functional status (Karnofsky score)" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.60, Regression, Cox — Unit of measure: Functional status (Karnofsky score). Functional status was estimated by the Karnofsky Performance Scale. Scores from 100 (Normal, no complaints) to 0 = (dead). 90 = Able to carry on normal activity. 80 = Normal activity with effort; Univariable Cox regression; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 2: Comparison: The Whole Study Group; The association of "Functional status (Karnofsky score 80 - 90 vs. 100)" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.48, Regression, Cox — Unit of measure: Functional status (Karnofsky score 80 - 90 vs. 100). Functional status was estimated by the Karnofsky Performance Scale (see Statistical analysis 1). P < 0.05 is regarded as statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.81 to 1.57]
Statistical Analysis 3: Comparison: The Whole Study Group; The association of "Functional status (Karnofsky score < 80 vs. 100)" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other — Univariable Cox regression; p = 0.63, Regression, Cox — Unit of measure: Functional status (Karnofsky score < 80 vs. 100). Functional status was estimated by the Karnofsky Performance Scale (see Statistical analysis 1). P < 0.05 is regarded as statistically significant; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.69 to 1.85]

26. Other Pre Specified Outcome: Analysis of the Social Factor "Visual Impairment" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline variable "Visual impairment" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 17 | 28 | 45
Statistical Analysis 1: Comparison: The Whole Study Group; The association of the Social Factor "Visual Impairment" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.71, Regression, Cox — Unit of measure: Visual impairment (yes vs. no). P-value < 0.05 is regarded as statistically significant; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.54 to 1.53]

27. Other Pre Specified Outcome: Analysis of the Social Factor "Impaired Hand Function" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Impaired hand function" (yes vs. no) in association with time to first peritonitis episode is presented. The impairment of hand function was unspecified. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 23 | 21 | 44
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Impaired Hand Function" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.29, Regression, Cox — Unit of measure: "Impaired Hand Function" (yes vs. no). P-value < 0.05 is considered statistically significant; Univariable Cox regression; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.80 to 2.06]

28. Other Pre Specified Outcome: Analysis of the Social Factor "Working Full or Part Time" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Working full or part time" (yes vs. no) in association with time to first peritonitis episode is presented.
  The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 103 | 102 | 205
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Working Full or Part Time" (yes vs. no) with time to first peritonitis episode analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.016, Regression, Cox — Units of measure: "Working full or part time (yes vs no)". P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.50 to 0.93]

29. Other Pre Specified Outcome: Analysis of the Social Factor "Retired" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Retired" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 184 | 169 | 353
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "being retired" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.041, Regression, Cox — Unit of measure: "Retired" (yes vs. no). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.01 to 1.73]

30. Other Pre Specified Outcome: Analysis of the Social Factor "Living Alone" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Living alone" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 91 | 77 | 168
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Living alone" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.064, Regression, Cox — Unit of measure: "Living alone" (yes vs. no). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.98 to 1.76]

31. Other Pre Specified Outcome: Analysis of the Social Factor "Need for Translation/Interpreter" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Working full or part time" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 9 | 13 | 22
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Need for translation/interpreter" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.14, Regression, Cox — Unit of measure: "Need for translation/interpreter" (yes vs. no). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.18 to 1.29]

32. Other Pre Specified Outcome: Analysis of the Social Factor "Current Smoking" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline social factor "Current smoking" (yes vs. no) in association with time to first peritonitis episode is presented. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 34 | 39 | 73
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Current smoking" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.60, Regression, Cox — Unit of measure: "Current smoking" (yes vs. no). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.75 to 1.65]

33. Other Pre Specified Outcome: Analysis of the Biochemical Characteristic "Serum Creatinine" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline biological characteristic Serum creatinine (micromol/L) in association with time to first peritonitis episode is presented. Serum creatinine was measured just before the start of peritoneal dialysis. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Micromol/L
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Micromol/L | 640 (234) | 650 (208) | 645 (222)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Serum creatinine (Hazard ratio per 100 micromol/L" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.18, Regression, Cox — Unit of measure: Serum creatinine (HR per 100 micromol/L". P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.90 to 1.02]

34. Other Pre Specified Outcome: Analysis of the Biochemical Characteristic "Serum Urea" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline biological characteristic Serum urea (mmol/L) in association with time to first peritonitis episode is presented. Serum urea was measured just before the start of peritoneal dialysis. The association of baseline variables (at PD start) with time to first peritonitis episode was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
mmol/L | 28 (9) | 28 (9) | 28 (9)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Serum urea (Hazard ratio per 5 mmol/l)" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.34, Regression, Cox — Unit of measure: Serum urea (Hazard ratio per 5 mmol/L). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.90 to 1.04]

35. Other Pre Specified Outcome: Analysis of the Biochemical Characteristic "Serum Albumin" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline biological characteristic" Serum albumin" (g/L) in association with time to first peritonitis episode is presented. Serum albumin was measured just before the start of peritoneal dialysis. The association of baseline variables (at PD start) with time to first peritonitis episode was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
g/L | 34 (6) | 34 (6) | 34 (6)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of Serum albumin (Hazard ratio per 5 g/L) with time to first peritonitis episode was analysed by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.019, Regression, Cox — Unit of measure: Serum albumin (Hazard ratio per 5g/L). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.79 to 0.98]

36. Other Pre Specified Outcome: Analysis of the Biochemical Characteristic "Serum Albumin (< 35 g/L vs. 35 g/L or More)" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline biological characteristic "Serum albumin" (< 35 g/L vs. 35 g/L or more) in association with time to first peritonitis episode is presented. Serum albumin was measured just before the start of peritoneal dialysis. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  Serum albumin <35 g/L | 169 | 169 | 338
  Serum albumin 35 g/L or more | 171 | 162 | 333
Statistical Analysis 1: Comparison: The Whole Study Group; Analysis of the association of serum albumin (<35 g/L vs. 35 g/l or more) with time to first peritonitis episode by univariable Cox regression. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.013, Regression, Cox — Unit of measure: Serum albumin (<35 g/L vs. 35 g/L or more). P-value <0.05 is regarded as significant; Univariable Cox regression; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.08 to 1.82]
Statistical Analysis 2: Comparison: The Whole Study Group; Analysis of the association of serum albumin (<35 g/L vs. 35 g/L or more) with time to first peritonitis episode by multivariable Cox regression; Test type: Other; p = 0.015, Regression, Cox — Unit of measure: Serum albumin (<35 g/l vs. 35 g/l or more). P-value <0.05 is regarded as significant; Multivariable Cox regression; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.06 to 1.82]

37. Other Pre Specified Outcome: Analysis of the Biochemical Characteristic "Haemoglobin" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of the baseline biological characteristic "Serum haemoglobin" (mmol/L) in association with time to first peritonitis episode is presented. Serum haemoglobin was measured just before the start of peritoneal dialysis. The association of baseline variables (at PD start) with time to first peritonitis was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
mmol/L | 110 (14) | 111 (12) | 111 (13)
Statistical Analysis 1: Comparison: The Whole Study Group; The association of Haemoglobin (Hazard ratio per 10 g/L) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.61, Regression, Cox — Unit of measure: Haemoglobin (HR per 10 g/L). P-value < 0.05 was considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.27 to 2.17]

38. Other Pre Specified Outcome: Analysis of the Use of a "Corticosteroid Drug" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The analysis of the use of a "Corticosteroid drug" (yes vs.no) in association with time to first peritonitis episode is presented. This variable may vary with time and is thus time-dependent. The variable was recorded at all study visits. The value recorded at the study visit which was closest to and prior to the first peritonitis episode was used in the univariable and multivariable Cox regression analyses of the association of the variable with time to first peritonitis episode. Time-dependent univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The count of participants on corticosteroid treatment at baseline is presented below.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 44 | 43 | 87
Statistical Analysis 1: Comparison: The Whole Study Group; The association of the time-dependent variable "Corticosteroid treatment" (yes vs. no) with time to first peritonitis episode was analysed by time-dependent univariable Cox regression; Test type: Other; p = 0.33, Regression, Cox — Unit of measure. The time-dependent variable "Corticosteroid treatment" (yes vs. no). Time-updated data were used. P-value < 0.05 was considered significant; Time-dependent univariable Cox regression; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.54 to 1.23]

39. Other Pre Specified Outcome: Analysis of "Cytotoxic Treatment" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: Analysis of "Cytotoxic treatment" (yes vs.no) in association with time to first peritonitis episode is presented. This variable may vary with time and is thus time-dependent. The variable was recorded at all study visits. The value recorded at the study visit which was closest to and prior to the first peritonitis episode was used in the time-dependent univariable and multivariable Cox regression analyses of the association of the variable with time to first peritonitis episode. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The count of participants on cytotoxic treatment at baseline is presented below.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 27 | 25 | 52
Statistical Analysis 1: Comparison: The Whole Study Group; The association of the time-dependent variable "Cytotoxic treatment" (yes vs. no) with time to first peritonitis episode was analysed by univariable time-dependent Cox regression; Test type: Other; p = 0.60, Regression, Cox — Unit of measure: Cytotoxic treatment (yes vs. no). Time-updated data was used. P-value < 0.05 was considered significant; Time-updated univariable Cox regression; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.70 to 1.84]

40. Other Pre Specified Outcome: Analysis of "Type of Start of Peritoneal Dialysis" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of "Type of start of peritoneal dialysis" in association with time to first peritonitis episode is presented. The type of start of peritoneal dialysis could be either planned or acute. The association of "Type of start of peritoneal dialysis" in association with time to first peritonitis episode was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  Planned PD start | 300 | 278 | 578
  Acute PD start | 40 | 53 | 93
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Type of PD start" with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.72, Regression, Cox — Unit of measure: Type of PD start (planned vs. acute). P-value < 0.05 was considered significant; Univariable Cox regression; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.73 to 1.57]

41. Other Pre Specified Outcome: Analysis of "The Use of Antibiotics Prior to PD Catheter Insertion" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The statistical analysis of "The use of antibiotics prior to PD catheter insertion" (yes vs. no) in association with time to first peritonitis episode is presented. Antibiotics prior to PD catheter insertion may be given to prevent infection. The association of "The use of antibiotics prior to PD catheter insertion" in association with time to first peritonitis episode was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The count of participants who used antibiotics prior to PD catheter insertion is presented below.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 305 | 305 | 610
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Antibiotics prior to PD catheter insertion" (yes vs. no) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.77, Regression, Cox — Unit of measure: Antibiotics prior to PD catheter insertion (yes vs. no). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.66 to 1.76]

42. Other Pre Specified Outcome: Analysis of "the Type of PD Catheter Used" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: PD catheters could be either be straight or coiled. The statistical analysis of "the type of PD catheter used" (straight vs. coiled) in association with time to first peritonitis episode is presented. The association of "the type of PD catheter used" in association with time to first peritonitis episode was studied in the whole study group. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  Straight PD catheter | 78 | 76 | 154
  Coiled PD catheter | 262 | 255 | 517
Statistical Analysis 1: Comparison: The Whole Study Group; The association of "Type of PD catheter used" (straight vs. coiled) with time to first peritonitis episode was analysed by univariable Cox regression; Test type: Other; p = 0.68, Regression, Cox — Unit of measure: Type of PD-catheter (straight vs. coiled). P-value < 0.05 is considered significant; Univariable Cox regression; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.68 to 1.28]

43. Other Pre Specified Outcome: Analysis of "PD Modality (CAPD/APD)" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: "PD modality (CAPD/APD)" in Association With Time to First Peritonitis Episode in the whole study group was studied. A participant either used CAPD (Continuous Ambulatory Peritoneal Dialysis) or APD (Automated Peritoneal Dialysis) but may change the PD modality during the study. This variable may vary with time and is thus time-dependent. The time-dependent data was recorded at all study visits. The value recorded at the study visit which was closest to and prior to the first peritonitis episode for each participant was used in the analyses. The time-dependent data was included in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The c
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants
  CAPD at PD start | 278 | 262 | 540
  APD at PD start | 62 | 69 | 131
Statistical Analysis 1: Comparison: The Whole Study Group; The PD modality (CAPD or APD) may vary with time and is thus time-dependent. Data were included as time-varying covariates in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the procedure was found; Test type: Other; p = 0.10, Regression, Cox — Unit of measure: PD modality (CAPD, continuous ambulatory peritoneal dialysis vs. APD, automated peritoneal dialysis). Time-updated data were used. P-value < 0.05 is regarded as significant; Univariable time-dependent Cox regression; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.96 to 1.66]

44. Other Pre Specified Outcome: Analysis of "Number of PD Bags Used/24h" in Association With of Time to First Peritonitis Episode in the Whole Study Group.
Description: The association of the "Number of PD bags used/24h" and Time to First Peritonitis Episode was studied. The number of PD bags used/24h many vary with time, as this variable is thus time-dependent. Data from PD start is presented below. As described in "Outcome measure 39", data was collected at each study visit. We recorded the number of bags connected to the PD catheter/24h in CAPD patients and in APD patients we recorded the number of bags connected to the tubing set/24h adding the daily number of bags connected to the PD catheter if additional manual daytime exchanges were used.
  The time-dependent data was included in a time-dependent univariable Cox regression to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: Number of PD bags/24h at PD start
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Number of PD bags/24h at PD start | 4 [1 to 5] | 4 [1 to 6] | 4. [1 to 6]
Statistical Analysis 1: Comparison: The Whole Study Group; The data regarding the number of PD bags used/24h were included as time-varying covariates in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity was found. The risk (hazard ratio) associated with the studied variable is reported; Test type: Other; p < 0.0001, Regression, Cox — Unit of measure: Number of PD bags used/24h. Time-updated data was used. P-value <0.05 was regarded as significant; Univariable time-dependent Cox regression. (The result of multivariable Cox regression is presented in Statistical analysis 2); Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.17 to 1.57]
Statistical Analysis 2: Comparison: The Whole Study Group; Analysis of the association of "Number of PD bags used per 24 hours with time to first peritonitis episode by multivariable time-dependent Cox regression. The multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with the studied variable is reported; Test type: Other; p < 0.0005, Regression, Cox — Unit of measure: Number of PD bags used /24h. Time-updated data was used. P-value < 0.05 was regarded as significant; Multivariable time-dependent Cox regression; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.13 to 1.54]

45. Other Pre Specified Outcome: Analysis of "The Volume of Dialysis Fluid Used/24h" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The association of "The Volume of Dialysis Fluid used/24h" with the time to first peritonitis episode is analysed in the whole study group. The volume of dialysis fluid used per 24h can vary with time and is thus time-dependent. The dialysis fluid volume/24h used at PD start is reported below. The time-dependent data were recorded at all study visits. The value recorded at the study visit, which was closest to and prior to the first peritonitis episode for each participant was used in the analyses. The time-dependent data were included in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: Liter of PD fluid used/24h at PD start
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Liter of PD fluid used/24h at PD start | 8.0 [1.5 to 18.5] | 8.0 [1.5 to 22.0] | 8.0 [1.5 to 22.0]
Statistical Analysis 1: Comparison: The Whole Study Group; Data regarding "Volume of dialysis fluid used/24h" was included as time-varying covariates in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity was found. The risk (hazard ratio) associated with the studied variable is reported; Test type: Other; p = 0.13, Regression, Cox — Unit of measure: Volume of dialysis fluid/24h (L). Time-updated data was used. P-value < 0.05 was considered significant; Univariable time-dependent Cox regression; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.99 to 1.08]

46. Other Pre Specified Outcome: Analysis of "Need of Help With Exit-site Care" in Association With Time to First Peritonitis Episode in the Whole Study Group.
Description: The exit site is the point where the PD catheter emerges from the skin of the abdomen. The number of "participants who needed of help with exit-site care at PD start is reported below. The need of this help may vary with time. This variable is thus time-dependent. The time-dependent data were recorded at all study visits. The value recorded at the study visit, which was closest to and prior to the first peritonitis episode for each participant was used in the analyses. The data were included as time-varying covariates in a time-dependent Cox regression. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 84 | 79 | 163
Statistical Analysis 1: Comparison: The Whole Study Group; Data regarding the variable "Help needed with exit-site care (yes vs. no)" were included as time-varying covariates in a univariable time-dependent Cox regression in order to identify variables significantly associated with time to first peritonitis episode. The risk (hazard ratio) associated with the studied variable is reported; Test type: Other; p = 0.79, Regression, Cox — Unit of measure: Help needed with exit-site care (yes vs. no). Time-updated data was used. P-value < 0.05 was considered significant; Univariable time-dependent Cox regression; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.77 to 1.41]

47. Other Pre Specified Outcome: Analysis of the Association of the Study Group (Retraining Group vs. the Control Group) With Time to First Peritonitis Episode
Description: Analysis of the association of the Study group (retraining group vs. control group) with time to first peritonitis episode is presented. Univariable Cox regression was used to identify variables significantly associated with time to first peritonitis episode. Multivariable Cox regression was performed using a backward elimination procedure stopping when all remaining factors were significant at p < 0.05. No collinearity among the factors affecting the backward elimination procedure was found. The risk (hazard ratio) associated with each studied variable is reported.
Time Frame: as for outcome 4
Population: 671 new patients with peritoneal dialysis (PD), peritonitis-free, aged 18 years or more, and able to perform PD without assistance were randomized to a control group and a retraining group.
Measure: Count of Participants; unit: Participants
Arm/Group | The Retraining Group | The Control Group | The Whole Study Group
Number analyzed (Participants) | 340 | 331 | 671
Participants | 340 | 331 | 671
Statistical Analysis 1: Comparison: The Retraining Group vs The Control Group; Association ot the Retraining group vs. the Control group with time to first peritonitis episode by univariable Cox regression; Test type: Other; p = 0.52, Regression, Cox — Unit of measure: Study group (retraining group vs. control group). P-value <0.05 is regarded as significant; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.71 to 1.19]

ADVERSE EVENTS:
Time Frame: The study participants were included from 18 Jan 2010 to 31 Dec 2014. They were followed up to 3 years. The study ended on 31 Dec 2015. No adverse events were reported in this study, which compared the number of peritonitis episodes which occurred in subjects with peritoneal dialysis who were given extra training in performing peritoneal dialysis and those who who were treated according the ordinary routines.
Description: No adverse events were expected in this kind of study and no adverse events were recorded.
Groups:
- The Follow-up Group: The intervention in the follow-up group consists of regular tests of the patients´ theoretical and practical skills regarding peritoneal dialysis. The test goals should be passed. If not, retraining will be given if needed til the goals are reached. The peritonitis rate in this group will be compared with that of the control group.
  Follow-up of PD patients´ theoretical and practical skills: Testing of patients knowledge and retraining if needed
Arm/Group | The Follow-up Group | Control Group
All-Cause Mortality (participants affected / at risk) | 27/340 | 29/331
Serious Adverse Events (participants affected / at risk) | 0/340 | 0/331
Other Adverse Events (participants affected / at risk) | 0/340 | 0/331

LIMITATIONS AND CAVEATS:
The limitations of the study mainly concerns its low power. The power calculation was based on a discontinuation rate of 30% of the participants after one year, However, 40% of the participants had left the study at that time. The power was also weakened by the fact that the recruitment to the study was slower than anticipated, and the final number of randomized participants was only 89% (671 0f 750) of the target, despite the fact that the inclusion time was extended from 2 years to 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No